CLINICAL TRIAL: NCT04165512
Title: Ultrasonographic Evaluation of the Effectiveness of Stellate Ganglion Block in Patients With Breast Cancer Related Lymphedema
Brief Title: Effectiveness of Stellate Ganglion Block in Breast Cancer Related Lymphedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09.2019.984
Record Dates: First submitted 2019-11-10; First posted 2019-11-18 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Lymphedema of Upper Limb; Breast Cancer Related Lymphedema
Keywords: lymphedema; breast cancer; stellate ganglion; treatment; ultrasound
MeSH Terms: conditions — Breast Cancer Lymphedema; Lymphedema; Breast Neoplasms | interventions — Bupivacaine; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stellate ganglion block in breast cancer related lymphedema (Experimental): US-guided stellat ganglion block will be applied to the patients with breast cancer related lymphedema twice at two-week intervals.
  Interventions: Combination Product: bupivacaine and triamcinolone

INTERVENTIONS:
Combination Product: bupivacaine and triamcinolone — a mixture of 4 mL 0.5% bupivacaine (marcaine) and 1 mL 40 mg triamcinolone (kenacort-a)
  Other Names: Marcaine; Kenacort-a

SUMMARY:
Lymphedema is a condition characterized by generalized or regional accumulation of protein-rich interstitial fluid as a result of impaired lymphatic circulation due to congenital or acquired disorders. Lymphedema is diagnosed through evaluations of its clinical criteria. Lymphedema is mostly evaluated through arm circumference measurements, water displacement measurements, tonometry, bioimpedance analysis, ultrasonography (US), computed tomography, lymphoscintigraphy and magnetic resonance imaging (MRI). Targets in the treatment of lymphedema include controlling the symptoms and preventing complications. A multimodal technique called complete decongestive therapy (CDT) is considered the gold standard of the treatment of lymphedema. In the literature, there are also studies showing that stellate ganglion block in breast cancer-related lymphedema treatment improves lymphedema and symptoms. Cervical stellate ganglion block is an invasive method used for the diagnosis and treatment of sympathetic pain and symptoms of upper extremity. Although it can be performed with fluoroscopy, CT and MRI, there has been increasing interest in ultrasound-guided technique since it has been fast, easy and cost-effective for the last few years. However, there are limited studies to provide sufficient evidence for the use of stellate ganglion block as an alternative treatment for lymphedema and detailed studies are needed in this area. The aim of this study is ultrasonographic evaluation of the efficacy of stellate ganglion block in the treatment of patients with breast cancer related lymphedema that is resistant to conservative treatment methods .

DETAILED DESCRIPTION:
Lymphedema is a condition characterized by generalized or regional accumulation of protein-rich interstitial fluid as a result of impaired lymphatic circulation due to congenital or acquired disorders. Lymphedema is diagnosed through evaluations of its clinical criteria. In addition to swelling of the affected extremities, certain symptoms, such as pain, fatigue, tightness, heaviness, tingling, weakness, and movement restriction, can also be seen in cases of lymphedema. Arm circumference measurements and volumetric methods are the most commonly used methods for calculating limb volume. In addition, soft tissue edema can be quantitatively measured by ultrasonography (US), computed tomography, lymphoscintigraphy and magnetic resonance imaging (MRI). Among these, US has been used more frequently in the evaluation of lymphedema. Ultrasonographic evaluation of the skin and subcutaneous tissue helps to determine the severity of lymphedema and the effectiveness of treatment. The reliability and utility of ultrasound in subcutaneous echogenicity grade (SEG) and subcutaneous echo-free space (SEFS) grade have been demonstrated in patients with breast cancer-related lymphedema. Targets in the treatment of lymphedema include controlling the symptoms and preventing complications. A multimodal technique called complete decongestive therapy (CDT) is considered the gold standard of the treatment of lymphedema. In the literature, there are also studies showing that stellate ganglion block in breast cancer-related lymphedema treatment improves lymphedema and symptoms. Cervical stellate ganglion block is an invasive method used for the diagnosis and treatment of sympathetic pain and symptoms of upper extremity. Although it can be performed with fluoroscopy, CT and MRI, there has been increasing interest in ultrasound-guided technique since it has been fast, easy and cost-effective for the last few years. However, there are limited studies to provide sufficient evidence for the use of stellate ganglion block as an alternative treatment for lymphedema and detailed studies are needed in this area. The aim of this study is ultrasonographic evaluation of the efficacy of stellate ganglion block in the treatment of patients with breast cancer related lymphedema that is resistant to conservative treatment methods.

Patients with breast cancer-related lymphedema will be evaluated for the study. For the diagnosis of lymphedema, detailed physical examination and limb circumference measurements will be performed. The patients with stage 2-3 lymphedema according to ISL staging, who had passed at least 3 months after breast surgery and did not response to conservative treatment methods will be included to the study. After obtaining written and oral informed consent of patients, US- guided stellate ganglion block will be applied two times at two-week intervals. Patients will be evaluated before injections (weeks 0 and 2) and 2 weeks after the last injection (week 4) and at 3 months of treatment. Arm circumference will be measured from 5 different areas, shoulder range of motion (ROM) will be evaluated with a goniometer, pain, and tightness and heaviness sensation will be assessed with visual analog scale. Quick-DASH questionnaire and Lymphedema Life Impcat scale will be applied to the patients. SEG and SEFS grade will be performed by evaluating subcutaneous tissue with USG.

After data collection, analysis will be performed with the appropriate statistical method.

ELIGIBILITY:
Inclusion Criteria:

* circumference difference of 2 cm or more between the affected and unaffected arm
* stage 2-3 lymphedema according to ISL staging
* aged between 18-70 years
* at least 3 months of follow-up breast surgery
* no response to the complete decongestive therapy enough

Exclusion Criteria:

* signs of cellulitis, lymphangitis, fungal infection,
* metastases to the lymph nodes
* uncontrolled psychiatric and systemic diseases
* contraindications for stellate ganglion block

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Arm circumference difference | before treatment (T0)
  Circumference differences between the affected and unaffected arms will be measured with a nonelastic tape measure at five levels; metacarpophalangeal joints, wrist, 15 cm distally from the medial epicondyle, medial epicondyle and 15 cm proximally from the medial epicondyle upper extremities.
Arm circumference difference | 2nd week of treatment (T1)
  Circumference differences between the affected and unaffected arms will be measured with a nonelastic tape measure at five levels; metacarpophalangeal joints, wrist, 15 cm distally from the medial epicondyle, medial epicondyle and 15 cm proximally from the medial epicondyle upper extremities.
Arm circumference difference | 4th week of treatment (T2)
  Circumference differences between the affected and unaffected arms will be measured with a nonelastic tape measure at five levels; metacarpophalangeal joints, wrist, 15 cm distally from the medial epicondyle, medial epicondyle and 15 cm proximally from the medial epicondyle upper extremities.
Arm circumference difference | 3rd month of treatment (T3)
  Circumference differences between the affected and unaffected arms will be measured with a nonelastic tape measure at five levels; metacarpophalangeal joints, wrist, 15 cm distally from the medial epicondyle, medial epicondyle and 15 cm proximally from the medial epicondyle upper extremities.
Subcutaneous echogenicity grade (SEG) | before treatment (T0)
  SEG will be performed by evaluating subcutaneous tissue with USG. Grade 0: No or little increase in echogenicity. Grade 1: Grade 1: Diffuse and monotonous increases in echogenicity Grade 2: Diffuse increases in echogenicity
Subcutaneous echogenicity grade (SEG) | 2nd week of treatment (T1)
  SEG will be performed by evaluating subcutaneous tissue with USG. Grade 0: No or little increase in echogenicity. Grade 1: Grade 1: Diffuse and monotonous increases in echogenicity Grade 2: Diffuse increases in echogenicity
Subcutaneous echogenicity grade (SEG) | 4th week of treatment (T2)
  SEG will be performed by evaluating subcutaneous tissue with USG. Grade 0: No or little increase in echogenicity. Grade 1: Grade 1: Diffuse and monotonous increases in echogenicity Grade 2: Diffuse increases in echogenicity
Subcutaneous echogenicity grade (SEG) | 3rd month of treatment (T3)
  SEG will be performed by evaluating subcutaneous tissue with USG. Grade 0: No or little increase in echogenicity. Grade 1: Grade 1: Diffuse and monotonous increases in echogenicity Grade 2: Diffuse increases in echogenicity
Subcutaneous echo-free space (SEFS) grade | before treatment (T0)
  SEFS grade will be performed by evaluating subcutaneous tissue with USG. Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (≥45 degrees to the skin) SEFS bridging the horizontally oriented SEFSs.
Subcutaneous echo-free space (SEFS) grade | 2nd week of treatment (T1)
  SEFS grade will be performed by evaluating subcutaneous tissue with USG. Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (≥45 degrees to the skin) SEFS bridging the horizontally oriented SEFSs.
Subcutaneous echo-free space (SEFS) grade | 4th week of treatment (T2)
  SEFS grade will be performed by evaluating subcutaneous tissue with USG. Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (≥45 degrees to the skin) SEFS bridging the horizontally oriented SEFSs.
Subcutaneous echo-free space (SEFS) grade | 3rd month of treatment (T3)
  SEFS grade will be performed by evaluating subcutaneous tissue with USG. Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (≥45 degrees to the skin) SEFS bridging the horizontally oriented SEFSs.
shoulder range of motion (ROM) will be evaluated with a goniometer | before treatment (T0)
  Shoulder range of motion (ROM) will be evaluated with a goniometer in all directions; flexion, extension, abduction, adduction, internal and external rotation.
shoulder range of motion (ROM) will be evaluated with a goniometer | 2nd week of treatment (T1)
  Shoulder range of motion (ROM) will be evaluated with a goniometer in all directions; flexion, extension, abduction, adduction, internal and external rotation.
shoulder range of motion (ROM) will be evaluated with a goniometer | 4th week of treatment (T2)
  Shoulder range of motion (ROM) will be evaluated with a goniometer in all directions; flexion, extension, abduction, adduction, internal and external rotation.
shoulder range of motion (ROM) will be evaluated with a goniometer | 3rd month of treatment (T3)
  Shoulder range of motion (ROM) will be evaluated with a goniometer in all directions; flexion, extension, abduction, adduction, internal and external rotation.
Pain, tightness and heaviness sensation | before treatment (T0)
  Shoulder pain and sensations of tightness and heaviness will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable)
Pain, tightness and heaviness sensation | 2nd week of treatment (T1)
  Shoulder pain and sensations of tightness and heaviness will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable)
Pain, tightness and heaviness sensation | 4th week of treatment (T2)
  Shoulder pain and sensations of tightness and heaviness will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable)
Pain, tightness and heaviness sensation | 3rd month of treatment (T3)
  Shoulder pain and sensations of tightness and heaviness will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable)

SECONDARY OUTCOMES:
Activity and participation - Quick-DASH | before treatment (T0)
  Quick-DASH is an assessment questionnaire that measures activity and participation limitations in all upper extremity disorders. The questionnaire assesses the difficulty of the daily life activities of the patients with 11 questions. Each answer is scored from 1 to 5 with a Likert scale. There is also two optional 4-item additional modules for whose jobs require a lot of upper limb performance and for sports people and musicians. The validity and reliability of the questionnaire in Turkish were conducted by Düger et al.
Activity and participation - Quick-DASH | 2nd week of treatment (T1)
  Quick-DASH is an assessment questionnaire that measures activity and participation limitations in all upper extremity disorders. The questionnaire assesses the difficulty of the daily life activities of the patients with 11 questions. Each answer is scored from 1 to 5 with a Likert scale. There is also two optional 4-item additional modules for whose jobs require a lot of upper limb performance and for sports people and musicians. The validity and reliability of the questionnaire in Turkish were conducted by Düger et al.
Activity and participation - Quick-DASH | 4th week of treatment (T2)
  Quick-DASH is an assessment questionnaire that measures activity and participation limitations in all upper extremity disorders. The questionnaire assesses the difficulty of the daily life activities of the patients with 11 questions. Each answer is scored from 1 to 5 with a Likert scale. There is also two optional 4-item additional modules for whose jobs require a lot of upper limb performance and for sports people and musicians. The validity and reliability of the questionnaire in Turkish were conducted by Düger et al.
Activity and participation - Quick-DASH | 3rd month of treatment (T3)
  Quick-DASH is an assessment questionnaire that measures activity and participation limitations in all upper extremity disorders. The questionnaire assesses the difficulty of the daily life activities of the patients with 11 questions. Each answer is scored from 1 to 5 with a Likert scale. There is also two optional 4-item additional modules for whose jobs require a lot of upper limb performance and for sports people and musicians. The validity and reliability of the questionnaire in Turkish were conducted by Düger et al.
Quality of life - Lymphedema Life Impact Scale | before treatment (T0)
  Lymphedema Life Impact Scale is a questionnaire developed to evaluate the physical, functional and psychosocial effects of lymphedema. It consists of 18 questions; It includes 8 physical, 4 psychosocial and 6 function subgroups. Each question is scored between 1 and 5, and high scores indicate increased severity. The validity and reliability of the Turkish version was made by Değirmenci et al.
Quality of life - Lymphedema Life Impact Scale | 2nd week of treatment (T1)
  Lymphedema Life Impact Scale is a questionnaire developed to evaluate the physical, functional and psychosocial effects of lymphedema. It consists of 18 questions; It includes 8 physical, 4 psychosocial and 6 function subgroups. Each question is scored between 1 and 5, and high scores indicate increased severity. The validity and reliability of the Turkish version was made by Değirmenci et al.
Quality of life - Lymphedema Life Impact Scale | 4th week of treatment (T2)
  Lymphedema Life Impact Scale is a questionnaire developed to evaluate the physical, functional and psychosocial effects of lymphedema. It consists of 18 questions; It includes 8 physical, 4 psychosocial and 6 function subgroups. Each question is scored between 1 and 5, and high scores indicate increased severity. The validity and reliability of the Turkish version was made by Değirmenci et al.
Quality of life - Lymphedema Life Impact Scale | 3rd month of treatment (T3)
  Lymphedema Life Impact Scale is a questionnaire developed to evaluate the physical, functional and psychosocial effects of lymphedema. It consists of 18 questions; It includes 8 physical, 4 psychosocial and 6 function subgroups. Each question is scored between 1 and 5, and high scores indicate increased severity. The validity and reliability of the Turkish version was made by Değirmenci et al.

CONTACTS AND LOCATIONS:
Overall Officials: Gülseren Akyüz, Prof, Study Chair — Marmara University; Canan Şanal-Toprak, Asst. Prof, Principal Investigator — Marmara University
Locations (1):
- Canan Şanal-Toprak, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suehiro K, Morikage N, Yamashita O, Harada T, Samura M, Takeuchi Y, Mizoguchi T, Nakamura K, Hamano K. Skin and Subcutaneous Tissue Ultrasonography Features in Breast Cancer-Related Lymphedema. Ann Vasc Dis. 2016;9(4):312-316. doi: 10.3400/avd.oa.16-00086. Epub 2016 Nov 25. PMID 28018504
- [Background] Kim J, Park HS, Cho SY, Baik HJ, Kim JH. The effect of stellate ganglion block on intractable lymphedema after breast cancer surgery. Korean J Pain. 2015 Jan;28(1):61-3. doi: 10.3344/kjp.2015.28.1.61. Epub 2015 Jan 2. PMID 25589949
- [Background] Kim JG, Bae SO, Seo KS. A comparison of the effectiveness of complex decongestive physiotherapy and stellate ganglion block with triamcinolone administration in breast cancer-related lymphedema patients. Support Care Cancer. 2015 Aug;23(8):2305-10. doi: 10.1007/s00520-014-2593-5. Epub 2015 Jan 11. PMID 25577504
- [Background] Park JH, Min YS, Chun SM, Seo KS. Effects of stellate ganglion block on breast cancer-related lymphedema: comparison of various injectates. Pain Physician. 2015 Jan-Feb;18(1):93-9. PMID 25675063
- [Background] Park MW, Lee SU, Kwon S, Seo KS. Comparison Between the Effectiveness of Complex Decongestive Therapy and Stellate Ganglion Block in Patients with Breast Cancer-Related Lymphedema: A Randomized Controlled Study. Pain Physician. 2019 May;22(3):255-263. PMID 31151333